CLINICAL TRIAL: NCT06339398
Title: Dose-response Effects of Physical Exercise Standardized Volume on Peripheral Biomarkers, Clinical Response and Brain Connectivity in Parkinson's Disease: a Prospective, Observational, Cohort Pilot Study
Brief Title: To Evaluate the Dose-response Effects of a Defined Volume of Physical Exercise on the Change of Peripheral Biomarkers, Clinical Response and Brain Connectivity in Parkinson's Disease: a Prospective, Observational, Cohort Pilot Study
Acronym: METEX-PD
Status: Recruiting | Type: Observational
Sponsor: Casa di Cura San Raffaele Cassino (Network)
Collaborators: IRCCS San Raffaele Roma (Other); San Raffaele Telematic University (Other); University of Rome Tor Vergata (Other); University of Urbino "Carlo Bo" (Other)
Responsible Party: Sponsor
Other Study IDs: 002-2023
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Physical exercise; Brain-derived neurotrophic factor (BDNF)
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Extensive Rehabilitation Group: PD patients of Extensive Group will perform a 45-minutes daily session of low-intensity aerobic exercise of 2-3 METs (37%-45% VO 2max ; 57-63% HR max) twice a week, for a 4-weeks period. Exercise volume: 180 METs-minutes/week
  Interventions: Behavioral: Aerobic exercise
- Intensive Rehabilitation Group: PD patients of Intensive Rehabilitation Group will exercise for 45 minutes daily at high-intensity aerobic training of 6-8.8 METs (46-91% VO2max ; 76-95% HRmax), five days per week, for 4-weeks period. Exercise volume:1350 METs-minutes/week
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Standardized volume of aerobic exercise, measured as METs-minutes/week

SUMMARY:
This is a prospective, observational, cohort pilot study of standardize volume of aerobic exercise on changes in BDNF concentration at 4-weeks of exercise training among Parkinson disease patients.

Thirty (N=30) participants will be consecutively enrolled and assigned to 2 groups: 1) Extensive Rehabilitation Group (exercise volume: 180 METs-min/week) or 2) Intensive Rehabilitation Group (exercise volume: 1350 METs-min/week).

The primary objective is to evaluate the dose-response effects of two different rehabilitation settings, characterized by different workload (measured as energy expenditure), on blood BDNF levels.

DETAILED DESCRIPTION:
This pilot observational study will evaluate the dose-response relationship between the volume of exercise, measured as METs-minutes/week, of two different rehabilitation settings to quantify the change in BDNF concentration in PD patients.

The study will also compare the changes induced by extensive and intensive rehabilitation settings in other neurotrophic factors and peripheral biomarkers, on motor and non-motor symptoms, kinematic parameters of gait, cognitive function, quality of life and the changes in cortical activity assessed with electroencephalogram (EEG) and in brain connectivity by functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease according to the United Kingdom (UK) Parkinson's Disease Society Brain Bank
* Aged between 30 and 80 years
* Disease stage II-III in "ON" phase according to modified Hoehn and Yahr (H&Y)
* Having no severe cognitive impairment:

  * Mini-Mental State Examination-MMSE ≥24
  * Montreal Cognitive Assessment - MoCA ≥ 17/30
* Under stable dopaminergic pharmacological treatment
* Motor condition that permits to execute 6-Minutes Walking Test (6MWT)
* Willing to participate in the study, understand the procedures and sign the informed consent.

Exclusion Criteria:

* Diagnosis of neurological disorders not related to Parkinson's disease
* Musculoskeletal diseases that could impair gait and execution of exercise program
* Presence of known cardiovascular disease that can compromise the performance required by the protocol
* Presence of diabetes or other metabolic and endocrine disease
* Uncontrolled hypertension (resting blood pressure >150/90 mmHg)
* Individuals with orthostatic hypotension and systolic pressure in feet below 100 will be excluded. Orthostatic hypotension (OH) is a reduction in systolic blood pressure of at least 20 mmHg or diastolic blood pressure of at least 10 mmHg within 3 minutes of standing.
* Hypo- or hyperthyroidism (TSH <0.5 or >5.0 mU/L), abnormal liver function (AST or ALT more than 2 times the upper limit of normal, ULN), alteration of kidney function.
* Values of complete blood test out of range and abnormal value clinically significant as per clinical judgment.
* Recent use of psychotropic drugs (e.g. anxiolytics, hypnotics, benzodiazepines, antidepressants) in which the dosage was not stable for 28 days before screening
* Severe disease (requiring systemic treatment and/or hospitalization) in the last 4 weeks.
* Any other clinically significant medical condition, psychiatric condition, drug or alcohol abuse, laboratory evaluation or abnormality that, in the opinion of the investigators, would interfere with the subject's ability to participate in the study.
* Beck Depression Inventory II (BDI) score > 28, indicating a severe depression that precludes the ability to exercise.
* (Only for women) State of pregnancy.
* Other disorders, injuries, diseases or conditions that may interfere with the ability to perform exercises (e.g. history of stroke, breathing problems, traumatic brain injury, orthopaedic injury or neuromuscular disease).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Brain-derived neurotrophic (BDNF) concentration assessed in peripheral blood samples (ng/mL) | 4 weeks
  Change from baseline (T0) in blood BDNF concentration
Change in Brain-derived neurotrophic (BDNF) concentration assessed in peripheral blood samples (ng/mL) | 8 weeks
  Change from baseline (T0) in blood BDNF concentration
Change in Brain-derived neurotrophic (BDNF) concentration assessed in peripheral blood samples (ng/mL) | 12 weeks
  Change from baseline (T0) in blood BDNF concentration

SECONDARY OUTCOMES:
Change in peripheral biomarker Insulin-like Growth Factor-1 (IGF-1) | 4 weeks
  Change from baseline (T0) in peripheral blood IGF-1 concentration (μg/L)
Change in peripheral biomarker Insulin-like Growth Factor-1 (IGF-1) | 8 weeks
  Change from baseline (T0) in peripheral blood IGF-1 concentration (μg/L)
Change in peripheral biomarker Insulin-like Growth Factor-1 (IGF-1) | 12 weeks
  Change from baseline (T0) in peripheral blood IGF-1 concentration (μg/L)
Change in peripheral biomarker Fibronectin type III domain-containing protein 5 (FNDC5)/Irisin | 4 weeks
  Change from baseline (T0) in FNDC5/Irisin by peripheral blood samples (ng/mL)
Change in peripheral biomarker Fibronectin type III domain-containing protein 5 (FNDC5)/Irisin | 8 weeks
  Change from baseline (T0) in FNDC5/Irisin by peripheral blood samples (ng/mL)
Change in peripheral biomarker Fibronectin type III domain-containing protein 5 (FNDC5)/Irisin | 12 weeks
  Change from baseline (T0) in FNDC5/Irisin by peripheral blood samples (ng/mL)
Change in peripheral biomarker of inflammation | 4 weeks
  Change from baseline (T0) in high sensitivity C-reactive protein (CRP) assessed by peripheral blood samples (mg/L)
Change in peripheral biomarker of inflammation | 8 weeks
  Change from baseline (T0) in high sensitivity C-reactive protein (CRP) assessed by peripheral blood samples (mg/L)
Change in peripheral biomarker of inflammation | 12 weeks
  Change from baseline (T0) in high sensitivity C-reactive protein (CRP) assessed by peripheral blood samples (mg/L)
Change in platelet distribution width (PDW) and number of platelets assessed by peripheral blood samples | 4 weeks
  Change from baseline (T0) in platelet distribution width (PDW) and number of platelets assessed by peripheral blood samples
Change in platelet distribution width (PDW) and number of platelets assessed by peripheral blood samples | 8 weeks
  Change from baseline (T0) in platelet distribution width (PDW) and number of platelets assessed by peripheral blood samples
Change in platelet distribution width (PDW) and number of platelets assessed by peripheral blood samples | 12 weeks
  Change from baseline (T0) in platelet distribution width (PDW) and number of platelets assessed by peripheral blood samples
Change in blood lactate levels assessed using finger-stick capillary blood samples | 4 weeks
  Change from baseline (T0) in blood lactate levels (mM) assessed using finger-stick capillary blood samples
Change in gut microbial diversity (species diversity %) assessed by next-generation sequencing (NGS) of the V3-V4 region of the 16S rDNA gene | 4 weeks
  Change from baseline (T0) in blood lactate levels (mM) assessed using finger-stick capillary blood samples
Change in motor symptoms - MDS-UPDRS part II | 4 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part II (motor symptoms of daily living). The minimum score on the MDS-UPDRS Part II is 0 and the maximum is 52 with higher scores representing worse motor symptoms of daily living
Change in motor symptoms - MDS-UPDRS part II | 8 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part II (motor symptoms of daily living). The minimum score on the MDS-UPDRS Part II is 0 and the maximum is 52 with higher scores representing worse motor symptoms of daily living
Change in motor symptoms - MDS-UPDRS part II | 12 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part II (motor symptoms of daily living). The minimum score on the MDS-UPDRS Part II is 0 and the maximum is 52 with higher scores representing worse motor symptoms of daily living
Change in motor symptoms - MDS-UPDRS part III | 4 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III (motor examination). The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132 with higher scores representing worse motor symptoms
Change in motor symptoms - MDS-UPDRS part III | 8 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III (motor examination). The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132 with higher scores representing worse motor symptoms
Change in motor symptoms - MDS-UPDRS part III | 12 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III (motor examination). The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132 with higher scores representing worse motor symptoms
Change in motor symptoms - MDS-UPDRS part IV | 4 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part IV (motor complication). The minimum score on the MDS-UPDRS Part IV is 0 and the maximum is 24 with higher scores representing worse motor complication
Change in motor symptoms - MDS-UPDRS part IV | 8 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part IV (motor complication). The minimum score on the MDS-UPDRS Part IV is 0 and the maximum is 24 with higher scores representing worse motor complication
Change in motor symptoms - MDS-UPDRS part IV | 12 weeks
  Change from baseline (T0) in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part IV (motor complication). The minimum score on the MDS-UPDRS Part IV is 0 and the maximum is 24 with higher scores representing worse motor complication
Change in movement analysis - stride length | 4 weeks
  Change from baseline (T0) in stride length [m], the distance between two consecutive hell strikes of the same foot evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - stride length | 8 weeks
  Change from baseline (T0) in stride length [m], the distance between two consecutive hell strikes of the same foot evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - stride length | 12 weeks
  Change from baseline (T0) in stride length [m], the distance between two consecutive hell strikes of the same foot evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - cadence | 4 weeks
  Change from baseline (T0) in cadence [steps/min], the number of steps in a minute evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - cadence | 8 weeks
  Change from baseline (T0) in cadence [steps/min], the number of steps in a minute evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - cadence | 12 weeks
  Change from baseline (T0) in cadence [steps/min], the number of steps in a minute evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - propulsion | 4 weeks
  Change from baseline (T0) in propulsion [m/ss], the anterior-posterior acceleration peak during the lower limb swing phase evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - propulsion | 8 weeks
  Change from baseline (T0) in propulsion [m/ss], the anterior-posterior acceleration peak during the lower limb swing phase evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - propulsion | 12 weeks
  Change from baseline (T0) in propulsion [m/ss], the anterior-posterior acceleration peak during the lower limb swing phase evaluated by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - Time Up and Go (TUG) | 4 weeks
  Change from baseline (T0) in execution timing of TUG, a reliable and valid test for assessing mobility, balance, walking ability and fall risk, by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - Time Up and Go (TUG) | 8 weeks
  Change from baseline (T0) in execution timing of Time Up and Go (TUG), a reliable and valid test for assessing mobility, balance, walking ability and fall risk, by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in movement analysis - Time Up and Go (TUG) | 12 weeks
  Change from baseline (T0) in execution timing of Time Up and Go (TUG), a reliable and valid test for assessing mobility, balance, walking ability and fall risk, by using a wearable device (G-sensor, BTS Bioengineering, Milan)
Change in walking capacity | 4 weeks
  Change from baseline (T0) in functional capacity evaluated by 6-minute Walking Test (6MWT), a standardized method to assess the maximal patient's capacity to walk as far as possible (measured in meters)
Change in walking capacity | 8 weeks
  Change from baseline (T0) in functional capacity evaluated by 6-minute Walking Test (6MWT), a standardized method to assess the maximal patient's capacity to walk as far as possible (measured in meters)
Change in walking capacity | 12 weeks
  Change from baseline (T0) in functional capacity evaluated by 6-minute Walking Test (6MWT), a standardized method to assess the maximal patient's capacity to walk as far as possible (measured in meters)
Change in postural instability | 4 weeks
  Change in Berg Balance Scale (BBS), which is a widely used clinical test to assess static and dynamic balance abilities
Change in postural instability | 8 weeks
  Change in Berg Balance Scale (BBS), which is a widely used clinical test to assess static and dynamic balance abilities
Change in postural instability | 12 weeks
  Change in Berg Balance Scale (BBS), which is a widely used clinical test to assess static and dynamic balance abilities
Change in cognitive function - Montreal Cognitive Assessment (MoCA) | 4 weeks
  Change from baseline (T0) in the MoCA. MoCA scores range between 0 and 30, with higher scores representing a better outcome
Change in cognitive function - Montreal Cognitive Assessment (MoCA) | 8 weeks
  Change from baseline (T0) in the MoCA. MoCA scores range between 0 and 30, with higher scores representing a better outcome
Change in cognitive function - Montreal Cognitive Assessment (MoCA) | 12 weeks
  Change from baseline (T0) in the MoCA. MoCA scores range between 0 and 30, with higher scores representing a better outcome
Change in cognitive function - Mini-Mental Examination (MMSE) | 4 weeks
  Change from baseline (T0) in the MMSE. MMSE scores range between 0 and 30, with higher scores representing a better outcome
Change in cognitive function | 8 weeks
  Change from baseline (T0) in the MMSE. MMSE scores range between 0 and 30, with higher scores representing a better outcome
Change in cognitive function | 12 weeks
  Change from baseline (T0) in the MMSE. MMSE scores range between 0 and 30, with higher scores representing a better outcome
Change in cognitive function - Frontal Assessment Battery (FAB) | 4 weeks
  Change from baseline (T0) in the FAB. FAB scores range between 0 and 18, with higher scores representing a better outcome
Change in cognitive function - Frontal Assessment Battery (FAB) | 8 weeks
  Change from baseline (T0) in the FAB. FAB scores range between 0 and 18, with higher scores representing a better outcome
Change in cognitive function - Frontal Assessment Battery (FAB) | 12 weeks
  Change from baseline (T0) in the FAB. FAB scores range between 0 and 18, with higher scores representing a better outcome
Change in severity of depressive symptomatology | 4 weeks
  Change from baseline (T0) in the Beck Depression Inventory-II (BDI-II).
Change in severity of depressive symptomatology | 8 weeks
  Change from baseline (T0) in the Beck Depression Inventory-II (BDI-II).
Change in severity of depressive symptomatology | 12 weeks
  Change from baseline (T0) in the Beck Depression Inventory-II (BDI-II).
Change in non-motor symptoms | 4 weeks
  Change from baseline (T0) in Non-Motor Symptoms Scale (NMSS) in PD
Change in non-motor symptoms | 8 weeks
  Change from baseline (T0) in Non-Motor Symptoms Scale (NMSS) in PD
Change in non-motor symptoms | 12 weeks
  Change from baseline (T0) in Non-Motor Symptoms Scale (NMSS) in PD
Change in motor fluctuations | 4 weeks
  Change from baseline (T0) in wearing OFF episodes will be assessed by Wearing OFF Questionnaire-19 (WOQ-19)
Change in motor fluctuations | 8 weeks
  Change from baseline (T0) in wearing OFF episodes will be assessed by Wearing OFF Questionnaire-19 (WOQ-19)
Change in motor fluctuations | 12 weeks
  Change from baseline (T0) in wearing OFF episodes will be assessed by Wearing OFF Questionnaire-19 (WOQ-19)
Change in quality of life | 4 weeks
  Change from baseline (T0) in will be measured with PDQ-39 questionnaire, which assesses how often PD patients experience difficulties across eight dimensions of daily living (0=never, 4=always).
Change in quality of life | 8 weeks
  Change from baseline (T0) in will be measured with PDQ-39 questionnaire, which assesses how often PD patients experience difficulties across eight dimensions of daily living (0=never, 4=always).
Change in quality of life | 12 weeks
  Change from baseline (T0) in will be measured with PDQ-39 questionnaire, which assesses how often PD patients experience difficulties across eight dimensions of daily living (0=never, 4=always).
Change in cortical activity | 4 weeks
  Change from the baseline (T0) in the cortical activity will be measured with resting-state electroencephalography (rsEEG)
Change in cortical activity | 12 weeks
  Change from the baseline (T0) in the cortical activity will be measured with resting-state electroencephalography (rsEEG)
Change in Brain Connectivity | 4 weeks
  Change from the baseline (T0) in brain connectivity through functional magnetic resonance imaging (fMRI).
Change in Brain Connectivity | 12 weeks
  Change from the baseline (T0) in brain connectivity through functional magnetic resonance imaging (fMRI).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Francesca De Pandis, MD,PhD, Principal Investigator — San Raffaele Cassino
Locations (1):
- San Raffaele Cassino, Cassino, Frosinone, Italy